CLINICAL TRIAL: NCT06294704
Title: Hybrid Closed Loop Insulin Pump and Bariatric Surgery in Patients With Type 1 Diabetes
Acronym: PompBariatDT1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0004
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery; Type 1 Diabetes
Keywords: Bariatric surgery; type 1 diabetes; hybrid closed-loop insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: bariatric surgery — Having undergone bariatric surgery and on a closed-loop insulin pump after bariatric surgery
  Other Names: Hybrid closed-loop insulin pump

SUMMARY:
Bariatric surgery is increasingly performed on patients with type 1 diabetes. It exposes these patients to an increased risk of hypoglycemia, including severe hypoglycemia, and of severe episodes of hyperglycemia, beyond the perioperative period. The long-term efficacy and safety of hybrid closed-loop insulin pump in these patients has not yet been published.

DETAILED DESCRIPTION:
Patients with type 1 diabetes and obesity are at risk of "double diabetes". Bariatric surgery may be indicated for these patients, to combat insulin resistance. Nevertheless, post-operative patients are at risk of hypoglycemia.

At the same time, patients with type 1 diabetes can benefit from a hybrid closed loop insulin pump to improve diabetes control and reduce the occurrence of hypoglycemia.

In type 1 diabetic patients who have undergone bariatric surgery and are treated with a hybrid closed loop insulin pump, continuous glucose measurement can be studied. In the medium and long term, the efficacy and safety of this system in this context will be described.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* With type 1 diabetes for > 1 year
* Obese (BMI≥30)
* Having undergone bariatric surgery
* On a hybrid closed-loop insulin pump
* Not pregnant
* No hybrid closed-loop insulin pump discontinuation for more than 45 days after surgery

Exclusion Criteria:

- Patient informed and opposed to data use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with type 1 diabetes who underwent bariatric surgery and treated by hybrid closed-loop insulin pump.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
time spent within glycemic target 70-180 mg/dL | at 3 months
  time spent within glycemic target 70-180 mg/dL in type 1 diabetes patients who underwent bariatric surgery,

SECONDARY OUTCOMES:
Time spent in level 1 hyperglycemia (181-250 mg/dL) | at 3 months
  Time spent in level 1 hyperglycemia (181-250 mg/dL)
  Time spent in level 1 hyperglycemia (181-250 mg/dL)
  Time spent in level 1 hyperglycemia (181-250 mg/dL)
Time spent in level 2 hyperglycemia (>250 mg/dL) | at 3 months
  Time spent in level 2 hyperglycemia (>250 mg/dL)
HbA1c | at 3 months
  HbA1c
Coefficient of variation | at 3 months
  Coefficient of variation
Time spent in level 1 hypoglycemia (51-70 mg/dl) | at 3 months
  Time spent in level 1 hypoglycemia (51-70 mg/dl)
Time spent in level 2 hypoglycemia (< 50 mg/gdl) | at 3 months
  Time spent in level 2 hypoglycemia (< 50 mg/gdl)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey BOULATE, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (3):
- France (3):
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France
  - CHU de Nantes, Nantes, France
  - APHP Hôpital de la Pitié Salpètrière, Paris, France

IPD SHARING:
Plan to Share IPD: No